CLINICAL TRIAL: NCT00261326
Title: Simvastatin Treatment of Patients With Acut Optic Neuritis. A Doubleblind, Randomized and Placebo Controlled Fase III Trial
Brief Title: Simvastatin Treatment of Patients With Acute Optic Neuritis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Collaborators: Alpharma ApS (Industry)
Responsible Party: MSci Jette Frederiksen, Glostrup Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Statin-01; KA 04068gs (Other: Regional scientific ethics Committe)
Record Dates: First submitted 2005-12-02; First posted 2005-12-05 (Estimated); Last update posted 2011-01-10 (Estimated); Status verified 2009-03

CONDITIONS: Optic Neuritis; Multiple Sclerosis
Keywords: Simvastatin; Optic Neuritis; Multiple Sclerosis
MeSH Terms: conditions — Optic Neuritis; Multiple Sclerosis | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B (Active Comparator): simvastatin tablets 80 mg daily
  Interventions: Drug: simvastatin
- A (Placebo Comparator): calcium tablets 80 mg
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: simvastatin — 80 mg once daily
  Arms: B
Drug: placebo — calcium tablets once daily
  Arms: A

SUMMARY:
The purpose of this study is to investigate if the simvastatin treatment improve the visual function after 3 months of the inclusion to this project and if the simvastatin influences the results on cerebral MRI after 3 and 6 months of the inclusion. In addition the development of new demyelinating relapses. In the patients with monosymptomatic acut optic neuritis to investigate whether the simvastatin reduces the risk to develop multiple sclerosis (MS).

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is a chronic inflammatory demyelinating disease in the Central Nervous System (CNS). Acute optic neuritis is a common symptom of MS and is considered to have the same pathogenesis as MS, where autoimmune and inflammatory mechanisms lead to the progression of MS.

Statins reduce the cholesterol in blood and in addition have anti-inflammatory effects. From experimental data and results from pilot projects there is evidence that the statins perform anti-inflammatory and immune-modulatory effects and one can expect a beneficial outcome in the autoimmune inflammatory diseases after the treatment with statins.

ELIGIBILITY:
Inclusion Criteria:

* Acute Optic Neuritis
* Abnormal contrast sensitivity score (>80)
* Symptom duration maximum 4 weeks
* Men and women between 18 and 59 years old
* The patient must be physical and mental able to participate i this project with a 6 months of the duration
* The patient must sign the written consent of the participation before the inclusion.

Exclusion Criteria:

* Optic neuritis earlier in the same eye
* Pregnancy
* Nursing
* Fertile women who do not use contraception
* Women who contemplate pregnancy in the duration of the study
* Steroid treatment the last 4 weeks before the inclusion
* Immune-supressor treatment the last 6 months before the inclusion
* Active liver disease or continuous increase of liver enzymes (ASAT, ALAT)without known reason.
* Kidney failure
* Myopathy
* Hyperthyroidism
* Diabetes mellitus
* Alcoholism
* Fibrates intake
* Statin treatment for other disease
* Simultaneous participation in other studies.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2006-09; Primary Completion 2010-01 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
The contrast sensibility of the eye after 3 months of the treatment | 6 months

SECONDARY OUTCOMES:
Visual acuity | 6 months
visual evokes potentials (VEP) | 6 months
cerebral MRI | 6 months
Developing MS after 6 months | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jette L Frederiksen, Dr.Med, Study Director
Locations (1):
- The clinic of the research for optic neuritis and MS, The Dpt. of Neurology at Glostrup Hospital, Glostrup Municipality, Glostrup, Denmark

REFERENCES:
- [Derived] Tsakiri A, Kallenbach K, Fuglo D, Wanscher B, Larsson H, Frederiksen J. Simvastatin improves final visual outcome in acute optic neuritis: a randomized study. Mult Scler. 2012 Jan;18(1):72-81. doi: 10.1177/1352458511415452. Epub 2011 Sep 15. PMID 21921071